CLINICAL TRIAL: NCT01838694
Title: Double-Blinded, Randomized, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Biochemical Activity of Intravenous Cpn10 Administration in Subjects With Mild to Moderate SLE.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Invion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IVXCpn001
Record Dates: First submitted 2013-04-17; First posted 2013-04-24 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Multiple doses of matched vehicle (no active ingredients) administered intravenously over 60 minutes.
  Interventions: Drug: Placebo
- Ala-Cpn10 (Experimental): Recombinant minimally modified Chaperonin10 (Cpn10) Multiple doses in the range 10mg twice weekly to 100mg twice weekly administered intravenously by infusion over 60 minutes.
  Interventions: Biological: Ala-Cpn10

INTERVENTIONS:
Biological: Ala-Cpn10
  Arms: Ala-Cpn10
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability, and efficacy of 4 weeks intravenous treatment with Cpn10 in subjects with mild to moderate active SLE.

ELIGIBILITY:
Inclusion Criteria (ALL must be met):

To be entered on study, subjects must meet the following criteria:

1. Male or female
2. Age 18 - 75 years
3. Patients fulfilling at least 4 criteria for SLE as defined by the American College of Rheumatology (ACR)
4. Laboratory values as follows:

   Documented ANA titer ≥ 1:160 or positive anti-dsDNA antibodies at, or any time prior to screening (verifiable laboratory result)
5. Not pregnant or breast-feeding
6. If corticosteroids are required for disease stability prior to study entry, able to tolerate a stable dose of ≤ 0.3 mg/kg/day of prednisone or equivalent for the duration of the study.
7. Agreement to use an effective form of contraception for the duration of the study.
8. Ability to understand and give consent.
9. Willing to participate and able to comply with the study requirements, procedures and visits.

   Mild SLE only
10. Present with mild active SLE disease

    Moderate SLE only
11. Present with active SLE disease based on SLE disease activity score (SLEDAI) ≥4 and ≤10
12. MCP-1 urinary level > 35 pg/ml
13. IL-6 serum level > 10 pg/ml
14. Meets the American College of Rheumatology (ACR) conditions for "renal disorder" as one of the diagnostic criteria for SLE i.e.

    1. Persistent proteinuria between 0.5 and 1.0 grams per day or > than 3+ by dipstick OR
    2. Cellular casts--may be red cell, hemoglobin, granular, tubular, or mixed

    OR
15. Physician (Pathologist) diagnosis of lupus nephritis of no greater severity than:

    1. Class I - Minimal mesangial lupus nephritis, OR
    2. Class II - Mesangial proliferative lupus nephritis, in accordance with the International Society of Nephrology (ISN) and the Renal Pathology Society (RPS) 2003 histological classification.

    With diagnosis made ≥ 6 months prior to study commencement.
16. If inclusion criteria #15 is met, subject must be receiving stable Standard of Care, including hydroxychloroquine, treatment appropriate for class I-II nephritis.

Exclusion Criteria (NONE can apply):

1. Active severe SLE flare with central nervous system (CNS) and/or renal manifestations, pericarditis, active pleuritis, active peritonitis or other SLE manifestations requiring treatment not allowed by the study protocol within 4 weeks of screening
2. Pregnant or breast-feeding
3. Lack of peripheral venous access.
4. History of cardiovascular disease. An acute cardiovascular event within 12 months of study entry, including arterial or venous thrombosis (blood clots).
5. Requirement for a stable dose of corticosteroid >0.3 mg/kg/day of prednisone or equivalent.
6. Active therapy with human or murine monoclonal antibodies (i.e. belimumab), within 2 months of study entry.
7. Any experimental therapy within 3 months of study entry.
8. Therapy with cyclophosphamide p.o or parenteral; pulse methylprednisolone or IVIG within 4-6 weeks.
9. Subjects being treated with sulfonylureas.
10. Subjects with any the following laboratory abnormalities: serum creatinine >3.0 mg/dL, WBC <3,500/μL, ANC <3,000/μL, absolute lymphocyte count ≤500/μL, Hgb <8.0 g/dL, platelets <50,000/μL, ALT and/or AST >1.5 x upper limit of normal (ULN), alkaline phosphatase >1.5 ULN.
11. Personal or psychiatric condition that precludes the subject being able to comply with the study requirements or understand and agree to the informed consent process.
12. Recent systemic bacterial, fungal, viral, or parasitic infections. Have required management/treatment or hospitalization for any infection within the last 4 weeks before screening.
13. History of malignancy - except completely excised basal cell carcinoma.
14. Impaired hepatic function
15. Body weight of 260lbs/120kg or more (BMI > 35)
16. History of tuberculosis (TB) or active, continuing treatment for TB
17. History of or current alcohol or substance abuse

    Mild SLE only
18. Active lupus nephritis and/or severe renal impairment (estimated or measured GFR < 50% predicted for age and gender)

    Moderate SLE only
19. Subjects with recently diagnosed lupus nephritis (diagnosis made <6 months prior to commencement of study
20. Subjects with active urinary sediment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Abel Buchheim Pharmaceutical Research, Miami, Florida
  - Northwestern University School of Medicine, Chicago, Illinois
  - Altoona Arthritis and Osteoporosis Center, Altoona, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Multiple doses of matched vehicle (no active ingredients) administered intravenously over 60 minutes.
  Placebo
- Ala-Cpn10: Recombinant minimally modified Chaperonin10 (Cpn10) Multiple doses in the range of 10mg twice weekly to 100mg twice weekly administered intravenously by infusion over 60 minutes.
  Ala-Cpn10
Period: Overall Study
Arm/Group | Placebo | Ala-Cpn10
Started | 8 | 22
Completed | 8 | 21
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ala-Cpn10 | Total
Number analyzed (Participants) | 8 | 22 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 18 | 24
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (18) | 43 (15) | 45 (15)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 21 | 28
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 22 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Serum Interleukin 6 (IL-6) Levels at the End of Active Dosing, Comparing Treatment to Placebo Cohort.
Time Frame: 4 weeks
Population: Analysis Population reflects participants for whom adequate analyzable samples were collected
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Ala-Cpn10 - 10mgs in Mild SLE: Recombinant minimally modified Chaperonin10 (Cpn10) 10mg twice weekly administered intravenously by infusion over 60 minutes.
  Ala-Cpn10
- Ala-Cpn10 - 30mgs in Mild SLE; Ala-Cpn10 - 30mgs in Moderate SLE: Recombinant minimally modified Chaperonin10 (Cpn10) 30mg twice weekly administered intravenously by infusion over 60 minutes.
  Ala-Cpn10
- Ala-Cpn10 - 100mgs in Mild SLE: Recombinant minimally modified Chaperonin10 (Cpn10) 100mg twice weekly administered intravenously by infusion over 60 minutes.
  Ala-Cpn10
Arm/Group | Placebo | Ala-Cpn10 - 10mgs in Mild SLE | Ala-Cpn10 - 30mgs in Mild SLE | Ala-Cpn10 - 100mgs in Mild SLE | Ala-Cpn10 - 30mgs in Moderate SLE
Number analyzed (Participants) | 5 | 5 | 4 | 3 | 1
percentage change from baseline | 1.6 (24.7) | 987.7 (2202.1) | -82.5 (20.4) | -29.7 (59.1) | 5000 (0)

ADVERSE EVENTS:
Time Frame: Up to 30 days following each patient's discontinuation of the study, for up to 9 weeks
Groups:
- Ala-Cpn10: Recombinant minimally modified Chaperonin10 (Cpn10) Multiple doses in the range (0.16mg/kg [10mg twice weekly] to 5mg/kg [300mg twice weekly]) administered intravenously by infusion over 60 minutes.
  Ala-Cpn10
Arm/Group | Placebo | Ala-Cpn10
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/22
Other Adverse Events (participants affected / at risk) | 4/8 | 6/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Ala-Cpn10 (N=22)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Ala-Cpn10 (N=22)
Eye pain (Eye disorders) | 1 | 0
diarrhoea (Gastrointestinal disorders) | 1 | 0
dyspepsia (Gastrointestinal disorders) | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3
Fatigue (General disorders) | 1 | 2
cutaneous lupus erythematosus (Immune system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less